CLINICAL TRIAL: NCT04734314
Title: Effect of Vojta on Balance and Quality of Life in Subject With Chronic Non-spacific Low Back Pain
Brief Title: Efficacy of Vojta on Balance and Quality of Life in Subject With CNLBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, walaa, principle investigator, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mtiu
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-04

CONDITIONS: Chronic Non-Specific Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment of back pain (Experimental): Group A: received conventional treatment of back pain which included; TENS 20 min and hot packs 10 min .The total treatment session is 30 min three session per week for four weeks
  Interventions: Other: conventional physical therapy
- vojta therapy (Experimental): received conventional treatment of back pain in addition to Vojta therapy . The total treatment session is 40 min.
  Interventions: Other: conventional physical therapy; Other: vojta therapy

INTERVENTIONS:
Other: conventional physical therapy — conventional physical therapy in the form of transcutaneous electrical stimulation (TENS) for 20 min and hot pack for 10 min Each patient received 12 sessions three session per week.
Other: vojta therapy — Vojta Dynamic Neuromuscular Stabilization (DNS) is a therapy used to manage neurological and musculoskeletal conditions each patient in the study group (group B) was instructed to lie prone on an examination table with the participant's shoulders abducted, elbows flexed approximately 80-90°, and the forearms hanging off the edge of the table. Pressure-like stimulation of the calcaneus and ASIS were performed in the postural position named by Vojta as "reflex creeping.
  Each patient received 12 sessions three session per week.
  Arms: vojta therapy

SUMMARY:
. To investigate the effect of Vojta method on static balance ,dynamic balance, quality of life in patients with chronic non - specific low back pain

DETAILED DESCRIPTION:
This randomized controlled trial is to investigate the effect of Vojta method on balance and quality of life in patients with chronic non-specific low back pain.

Forty patients (male and female) complaining of chronic non -specific low back pain was recruited to share in this study

. The recruited patients were randomly recruited into two groups; group A (control group) and group B (study group).

Group A: received conventional treatment of back pain which included; TENS 20 min and hot packs 10 min .The total treatment session is 30 min three session per week for four weeks Group B: received conventional treatment of back pain in addition to Vojta method. The total treatment session is 40 min.

Patient in both groups performed 10 sessions, 3 session per week

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic non -specific low back pain for more than 3 months.
2. Their age ranged between 18-35 years old
3. Both sexes were recruited in this study.
4. Their BMI ranged between 18-25 kg/m2

Exclusion Criteria:

1- Patients with previous spinal surgery 2. Patients who have radiological diagnosis of spondylolysis or spondylolisthesis.

3. Patient with neurological disease . 4. Chest problems 5. Systematic disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-02-05 (Estimated); Study Completion 2021-02-05 (Estimated)

PRIMARY OUTCOMES:
static and dynamic balance | one month
  static and dynamic balance can assessed by using biodex balance system Each patient was instructed to maintain his/her balance for the period of the test.
  There was report gained after finishing every test includes information on medial lateral stability index(MLSI), overall stability index(OSI), and anterior posterior stability index (APSI) measurements will done twice before and after treatment for all patients in both group
Oswestry Low Back Pain Disability Questionnaire | one month
  The Oswestry Low Back Pain Disability Questionnaire is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability and quality of life. The test is considered the 'gold standard' of low back functional outcome tools measurements will done twice before and after treatment for all patients in both group

CONTACTS AND LOCATIONS:
Locations (1):
- Mti University, Cairo, Egypt